CLINICAL TRIAL: NCT06651333
Title: Functional Connectivity Mechanisms of Opioid Abstinence
Brief Title: fMRI and Opioid Abstinence
Status: Recruiting | Type: Observational
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2000038046; 1R01DA060631-01 (NIH)
Record Dates: First submitted 2024-10-18; First posted 2024-10-21 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Drug Use Disorder; Opioid Dependence; Opioid-Related Disorders; Opioid Use; Opioid Abuse
Keywords: Relapse
MeSH Terms: conditions — Substance-Related Disorders; Opioid-Related Disorders; Recurrence | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Methadone: Participants initiated into methadone within the past 6 months will receive fMRI and cognitive assessment battery.
  Interventions: Diagnostic Test: fMRI
- Buprenorphrine: Participants initiated into buprenorphine within the past 6 months will receive fMRI and cognitive assessment battery.
  Interventions: Diagnostic Test: fMRI

INTERVENTIONS:
Diagnostic Test: fMRI — Participants will be performing tasks while undergoing fMRI. Tasks include Stroop task, Emotion-regulation task and an Ambiguity reward task, Drug cue task, and Cognitive behavioral therapy task. Participants are not presented with any specific stimulus.

SUMMARY:
This project examines functional connectivity patterns associated with subsequent relapse to illicit opioids during treatment for OUD.

ELIGIBILITY:
Inclusion Criteria:

* recent initiation of methadone or buprenorphine at a clinic or program within the past year (i.e., period of time during which treatment drop-out and risk for relapse is highest);
* eligibility for MRI scanning;
* ability to commit to study visits.

Exclusion Criteria:

* current acute psychosis, mania, or suicidal ideation with intent, as assessed during screening with the SCID-5;
* current intoxication or acute withdrawal at time of study visit sufficient to prevent participation based on: behavioral observation, breathalyzer, and SOWS assessment;
* severe cognitive impairment as determined via trained clinical research staff through consent process and during consent quiz or as indicated by a PROMIS Cognitive Function tscore <30 (i.e., severe impairment)
* past or present history of intellectual disability, developmental disorder, or neurological disease;
* head trauma with loss of consciousness >30 min;
* organ dysfunction or any unstable or untreated medical conditions that may interfere with study participation.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Participants will be individuals with primary opioid use disorder who are at least 18 years old and enrolled in formal MOUD treatment (either methadone or buprenorphine) for less than 6 months. Investigators will recruit a sample that is 50% female and 50% male.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2029-11 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Illicit opioid-use | At monthly visits for 6 months following neuroimaging
  Defined as the percent days of self-reported use of illicit opioids (assessed at monthly visits for 6-months following neuroimaging), with the exception of primary type of MOUD (i.e., methadone for methadone treated individuals, buprenorphine for buprenorphine treated individuals).

SECONDARY OUTCOMES:
MOUD retention | up to 9 months
  Percentage of visits attended out of visits expected based on electronic health record data and time line follow back.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Yip, PhD, MSc, Principal Investigator — Yale University
Locations (1):
- The APT Foundation, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
This study will submit and share data with OpenNeuro. This will include de-identified demographic data, neuropsychological assessment data, clinical assessment data, and fMRI data (raw).
Time Frame: All data will be deposited to OpenNeuro starting 24 months after data collection begins and will be deposited every six months thereafter. OpenNeuro policy states that any data uploaded to their repository becomes publicly available under a Creative Commons CC0 license after a 36-month period beginning from first successful version of the dataset.
Access Criteria: OpenNeuro policy states that any data uploaded to their repository becomes publicly available under a Creative Commons (CC) license after a 36-month period beginning from first successful version of the dataset. Users create an account with OpenNeuro account in order to download BIDS formatted files and any associated metadata.